CLINICAL TRIAL: NCT05621200
Title: Interventional Cross-over Study to Evaluate the Efficacy on Motor and Cognitive Performance of Transcranial Alternating Current Stimulation (tACS) in Patients With Neurodegenerative Ataxia
Brief Title: Transcranial Alternating Current Stimulation (tACS) in Patients With Ataxia
Acronym: SCAtACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NP4514
Record Dates: First submitted 2022-10-20; First posted 2022-11-17 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Ataxia; Spinocerebellar Ataxias; Multiple System Atrophy; Ataxia With Oculomotor Apraxia; CANVAS
Keywords: transcranial direct current stimulation; transcranial alternate current stimulation; spinocerebellar ataxia; cerebellar ataxia
MeSH Terms: conditions — Ataxia; Spinocerebellar Ataxias; Multiple System Atrophy; Spinocerebellar ataxia, autosomal recessive 1; Cerebellar Ataxia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transcranial direct current stimulation (tDCS) (Active Comparator): Single session of anodal tDCS at 2 mA over the cerebellar hemispheres
  Interventions: Device: Transcranial stimulation over the cerebellar hemispheres
- Transcranial alternate current stimulation (tDCS) (Active Comparator): Single session of gamma tACS (50 Hz) at 3 mA over the cerebellar hemispheres
  Interventions: Device: Transcranial stimulation over the cerebellar hemispheres
- Placebo stimulation (sham) (Sham Comparator): Single session of sham tDCS over the cerebellar hemispheres
  Interventions: Device: Transcranial stimulation over the cerebellar hemispheres

INTERVENTIONS:
Device: Transcranial stimulation over the cerebellar hemispheres — Single session of Transcranial stimulation over the cerebellar hemispheres

SUMMARY:
The aim of the study is to evaluate the effects on motor and cognitive performance of transcranial alternating current stimulation (tACS) compared to transcranial direct current stimulation (tDCS) and placebo stimulation (sham) in patients with neurodegenerative ataxia to identify a possible rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cerebellar syndrome and quantifiable cerebellar atrophy

Exclusion Criteria:

* Severe head trauma in the past
* History of seizures
* History of ischemic stroke or hemorrhage
* Pacemaker
* Metal implants in the head/neck region
* Severe comorbidity
* Intake of illegal drugs
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change in the International Cooperative Ataxia Rating Scale (ICARS) Score From Baseline | Baseline (immediately before the intervention) - Immediately after the intervention
  International Cooperative Ataxia Rating Scale (ICARS): semi-quantitative 100-point scale, yielding a total score of 0 (no ataxia) to 100 (most severe ataxia).
Change in the Scale for the Assessment and Rating of Ataxia (SARA) Score From Baseline | Baseline (immediately before the intervention) - Immediately after the intervention
  Scale for the Assessment and Rating of Ataxia (SARA): 8-item performance based scale, yielding a total score of 0 (no ataxia) to 40 (most severe ataxia).

SECONDARY OUTCOMES:
Change in Cerebellar Brain Inhibition (CBI) Measurements From Baseline | Baseline (immediately before the intervention) - Immediately after the intervention
  Cerebellar brain inhibition (CBI) is expressed as motor evoked potential amplitude (average of 10 recordings). Lower values reflect higher inhibition and thus reduced impairment.
Change in Timed Up and Go Test Duration From Baseline | Baseline (immediately before the intervention) - Immediately after the intervention
  Time (in seconds) that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees, assessed with gait sensors.
Change in Walking Cadence From Baseline | Baseline (immediately before the intervention) - Immediately after the intervention
  Average Left and Right Steps/Minute during a 60 seconds walk, assessed with gait sensors.
Change in 360° Turn From Baseline | Baseline (immediately before the intervention) - Immediately after the intervention
  Velocity (Number of Degrees/sec) in making a 360° turn, assessed with gait sensors

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Borroni, MD, Principal Investigator — ASST Spedali Civili di Brescia; Alberto Benussi, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benussi A, Dell'Era V, Cantoni V, Bonetta E, Grasso R, Manenti R, Cotelli M, Padovani A, Borroni B. Cerebello-spinal tDCS in ataxia: A randomized, double-blind, sham-controlled, crossover trial. Neurology. 2018 Sep 18;91(12):e1090-e1101. doi: 10.1212/WNL.0000000000006210. Epub 2018 Aug 22. PMID 30135258
- [Background] Benussi A, Dell'Era V, Cotelli MS, Turla M, Casali C, Padovani A, Borroni B. Long term clinical and neurophysiological effects of cerebellar transcranial direct current stimulation in patients with neurodegenerative ataxia. Brain Stimul. 2017 Mar-Apr;10(2):242-250. doi: 10.1016/j.brs.2016.11.001. Epub 2016 Nov 3. PMID 27838276
- [Background] Benussi A, Koch G, Cotelli M, Padovani A, Borroni B. Cerebellar transcranial direct current stimulation in patients with ataxia: A double-blind, randomized, sham-controlled study. Mov Disord. 2015 Oct;30(12):1701-5. doi: 10.1002/mds.26356. Epub 2015 Aug 14. PMID 26274840
- [Background] Benussi A, Cantoni V, Manes M, Libri I, Dell'Era V, Datta A, Thomas C, Ferrari C, Di Fonzo A, Fancellu R, Grassi M, Brusco A, Alberici A, Borroni B. Motor and cognitive outcomes of cerebello-spinal stimulation in neurodegenerative ataxia. Brain. 2021 Sep 4;144(8):2310-2321. doi: 10.1093/brain/awab157. PMID 33950222
- [Derived] Libri I, Cantoni V, Benussi A, Rivolta J, Ferrari C, Fancellu R, Synofzik M, Alberici A, Padovani A, Borroni B. Comparing Cerebellar tDCS and Cerebellar tACS in Neurodegenerative Ataxias Using Wearable Sensors: A Randomized, Double-Blind, Sham-Controlled, Triple-Crossover Trial. Cerebellum. 2024 Apr;23(2):570-578. doi: 10.1007/s12311-023-01578-6. Epub 2023 Jun 22. PMID 37349632